CLINICAL TRIAL: NCT05805007
Title: A Single-arm, Open-label Exploratory Clinical Study to Assess the Preliminary Safety of the Gene Editing Drug ZVS203e for the Management of Retinitis Pigmentosa Caused by Mutations in the RHO Gene
Brief Title: Safety and Tolerability Study of Gene Editing Drug ZVS203e in Participants With Retinitis Pigmentosa
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYB-2022-001
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Retinitis Pigmentosa
Keywords: gene editing; retinitis pigmentosa; RHO; rAAV
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): Three cohorts of 3 patients each. All the patients enrolled in the study will receive a single subretinal injection in one eye.
  Cohort 1: Subretinal administration of a single low dose ZVS203e at Day 0. Cohort 2: Subretinal administration of a single medium dose ZVS203e at Day 0. Cohort 3: Subretinal administration of a single high dose ZVS203e at Day 0.
  Interventions: Drug: ZVS203e

INTERVENTIONS:
Drug: ZVS203e — ZVS203e is a rAAV-mediated gene editing drug that silences RHO mutant protein expression by CRISPR/Cas9 editing system.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of a single escalating doses of ZVS203e administered via subretinal injection in participants with RP caused by RHO site-specific gene mutation (RHO-RP).

DETAILED DESCRIPTION:
This is a single-arm, open-label, single ascending dose study of ZVS203e in participants with RHO-RP. Up to 9 participants will be enrolled in this study. Safety, efficacy and vector shedding characteristics of ZVS203e are then measured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with clinical diagnosis of Retinitis Pigmentosa (RP) (age ≥ 18 years) ;
* 2. Genetic test confirmed to carry a fix mutation of RHO and carry no pathogenic mutations of other ophthalmic genetic diseases;
* 3. Meet the following target eye selection criteria： Best corrected visual acuity between 2.3 LogMAR and 0.5 LogMAR (including 2.3 LogMAR and 0.5 LogMAR, equivalent to Snellen visual acuity of hand move to 20/63) ;
* 4. Agree to take effective contraceptive measures from the beginning of the study to 1 year after the administration;
* 5.Willingness to adhere to protocol as evidenced by written informed consent;

Exclusion Criteria:

* 1. Existing or pre-existing of macular lesions such as retinoschisis or macular membrane, or other eye conditions interfering with the surgery or the interpretation of the clinical endpoint, in the investigators' opinion;
* 2. The study eye has been treated with other drugs within 3 months that could affect the evaluation of the investigational drug;
* 3. The study eye has been treated with the following intraocular procedures: retinal detachment surgery, vitrectomy;
* 4. The presence of an ocular/visual disease, disorder or lesion known to cause, or to be associated with, vision loss, or whose associated treatment or therapy is known to cause, or to be associated with, vision loss；
* 5. Currently taking or may require systemic medications that can cause ocular toxicity, such as psoralen, risedronate, or tamoxifen;
* 6. Known allergy to the drug planned for use in the study；
* 7.Those with the following laboratory abnormalities which are clinically significant: Liver function: chronic liver disease, ALT increased >2 times the upper limit of normal; With uncontrolled hypertension, mean systolic blood pressure ≥ 160 mmHg or mean diastolic blood pressure ≥ 100 mmHg; With uncontrolled diabetes, HbA1c>10%; Patients with abnormal coagulation function (prothrombin time ≥ upper limit of normal (3 seconds' longer), activated partial thromboplastin time ≥ upper limit of normal (10 seconds' longer)); Serum virology test: Active hepatitis B, hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) or syphilis antibody positive;
* 8. Having any past or present medical history that may affect the safety of the trial or the in vivo process of the drug, especially the medical history of cardiovascular, hepatic, renal, endocrine, gastrointestinal, pulmonary, neurological, hematological, oncologic, immunological or metabolic disorders and others that are thought clinically significant by the investigator；
* 9. Participation in any medicine or medical device clinical trials within 3 months prior to enrollment;
* 10. Neutralizing antibodies to rAAV> 1:1000 by immunologic test;
* 11. For females in pregnancy or lactation period;
* 12. Any other conditions which leads the investigator to determine the participant is unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs） | Baseline up to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events (SAEs) | Baseline up to Week 52
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that leading to the following:
  Results in death; Life-threatening, refers to an event in which the patient is at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe; Significant or permanent disability/incapacity, where disability refers to a serious disruption and damage of a person's ability to perform normal life functions; Requires inpatient hospitalization or prolongation of existing hospitalization; Congenital anomaly or birth defect; Other medically important events.

SECONDARY OUTCOMES:
Mean change from baseline in BCVA after ZVS203e treatment | Baseline up to Week 52
  BCVA of both eyes will be assessed using the early treatment of diabetic retinopathy study (ETDRS) chart.
Change from Baseline in visual field | Baseline up to Week 52
  Visual field will be assessed by Humphrey perimetry, changes in VFI, MD, PSD will be analyzed.
Change from Baseline in contrast sensitivity | Baseline up to Week 52
  Change from baseline in contrast sensitivity will be measured using the CSV-1000E instrument.
Change from Baseline in multi-luminance mobility test (MLMT) | Baseline up to Week 52
  MLMT was assessed at 1 or more of 7 levels of illumination, ranging from 400 lux (a brightly lit office) to 1 lux (a moonless summer night). The score range is between -1 (the worst) and 6 (the best).
Change from Baseline in retinal thickness | Baseline up to Week 52
  Retinal thickness will be assessed for both eyes using OCT.
Change from Baseline in fundus autofluorescence (FAF) | Baseline up to Week 52
  FAF is a noninvasive test to explore the health and metabolic status of retinal pigment epithelial cell/photoreceptor complex.
Change from Baseline in color vision | Baseline up to Week 52
  Subjects' color vision was classified and graded by Farnsworth Munsell 100 hue.
Change from Baseline in mfERG | Baseline up to Week 52
  The measurement will be performed based on the standards of international society for clinical electrophysiology of vision (ISCEV).
Change from Baseline in NEI VFQ-25 total score | Baseline up to Week 52
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Liping Yang, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No